CLINICAL TRIAL: NCT07186504
Title: Impact of Adapted Physical Activity Combined With Pelvic Floor Functionality on Pelvic Girdle Pain During Pregnancy: A Randomized Controlled Exploratory Trial
Brief Title: Adapted Physical Activity and Pelvic Floor Function for Pelvic Girdle Pain During Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: La Tour Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01561
Record Dates: First submitted 2025-09-01; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Girdle Pain; Pregnancy; Pelvic Floor Dysfunctions
Keywords: Pregnancy-related pelvic girdle pain; Prenatal pelvic pain; Pelvic floor function; Pelvic floor rehabilitation; Adapted physical activity; Prenatal exercise; Physiotherapy in pregnancy; Prenatal musculoskeletal pain; Maternal health; Randomized controlled trial
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a monocentric, randomized, controlled, open-label exploratory trial with two parallel arms. Forty pregnant women with clinically confirmed pelvic girdle pain will be randomized (1:1) to an intervention group or a control group. The intervention group will participate in weekly sessions of adapted physical activity, specifically designed for pregnant women with pelvic girdle pain, until 36-38 weeks of gestation. If pelvic floor dysfunction is identified, individualized pelvic floor rehabilitation will be added. The control group will receive standard prenatal care and a flyer with international recommendations on safe physical activity during pregnancy. Outcomes will be assessed at baseline (≤27 weeks of gestation), late pregnancy (36-38 weeks), and 3 months postpartum.
Masking Description: This is an open-label trial. Neither participants nor investigators are blinded to group assignment due to the nature of the intervention (supervised physical activity and rehabilitation). Outcome assessments are self-reported or clinician-administered and not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity with or without Pelvic Floor Rehabilitation (Experimental): Participants attend weekly 60-minute sessions of adapted physical activity, from enrollment (≤27 weeks gestation) until 36-38 weeks of pregnancy. Sessions alternate between land and aquatic settings and include mobility, lumbopelvic stabilization, core and multifidus strengthening, and safe aerobic training. If pelvic floor dysfunction is identified at baseline using the Pelvic Floor Distress Inventory (PFDI-20), participants will also receive individualized pelvic floor rehabilitation (up to 9 sessions) focusing on pelvic floor muscle relaxation, strengthening, and coordination.
  Interventions: Behavioral: Adapted Physical Activity; Behavioral: Pelvic Floor Rehabilitation
- Standard Care and Educational Flyer (Active Comparator): Participants receive standard prenatal care as provided by their healthcare providers. In addition, they are given a validated flyer containing international recommendations for safe physical activity during pregnancy. No supervised physiotherapy or structured exercise sessions are provided.
  Interventions: Other: Standard Care (in control arm); Other: Educational Flyer

INTERVENTIONS:
Behavioral: Adapted Physical Activity — Group-based, weekly supervised 60-minute sessions including mobility, stability, strengthening, and aerobic exercises adapted for pregnancy and pelvic girdle pain.
  Arms: Adapted Physical Activity with or without Pelvic Floor Rehabilitation
Behavioral: Pelvic Floor Rehabilitation — Individual physiotherapy sessions using the PERFECT scheme to assess and retrain pelvic floor muscle function, including education, manual therapy, relaxation, and strengthening
  Arms: Adapted Physical Activity with or without Pelvic Floor Rehabilitation
Other: Standard Care (in control arm) — Usual prenatal care provided by obstetricians or midwives according to local practice.
  Arms: Standard Care and Educational Flyer
Other: Educational Flyer — Written information with evidence-based international guidelines on physical activity during pregnancy.
  Arms: Standard Care and Educational Flyer

SUMMARY:
Pelvic girdle pain (PGP) is a common condition during pregnancy, affecting up to two-thirds of women. It can cause significant discomfort, limit daily activities, and reduce quality of life. Current treatment options are limited, and many women continue to experience pain throughout pregnancy and even after childbirth.

This study will evaluate whether a structured program of adapted physical activity, with additional individualized pelvic floor rehabilitation when needed, can reduce pelvic girdle pain and improve function during pregnancy. The intervention consists of weekly 60-minute sessions of adapted physical activity, led by a pelvic health physiotherapist, from inclusion until 36-38 weeks of gestation. The exercises focus on lumbopelvic stability, mobility, strengthening, and safe aerobic activity. If a participant presents with pelvic floor dysfunction, individualized rehabilitation may be added in parallel.

Participants will be randomly assigned to either the intervention group (adapted physical activity ± pelvic floor rehabilitation) or a control group. The control group will receive standard pregnancy follow-up care plus a validated flyer with international recommendations on physical activity during pregnancy but without supervised sessions.

The primary outcomes are pain intensity and functional impact of PGP, measured using the Visual Analog Scale (VAS) and the Pelvic Girdle Questionnaire (PGQ). Secondary outcomes include self-reported physical activity, pelvic symptoms, pelvic floor function, adherence to the intervention, and acceptability of the program.

A total of 40 pregnant women will be enrolled at Hospital La Tour in Geneva, Switzerland. Assessments will take place at three time points: inclusion (≤27 weeks of gestation), late pregnancy (36-38 weeks), and 3 months after delivery.

The study is expected to provide new evidence on the benefits of integrating pelvic floor functionality into physical activity programs for pregnant women with PGP. If effective, this approach could inform clinical practice and improve care for women during pregnancy

DETAILED DESCRIPTION:
Background and Rationale

Pregnancy induces substantial morphological, hormonal, and biomechanical changes that increase the risk of musculoskeletal pain, particularly pelvic girdle pain (PGP). Up to 63% of pregnant women experience PGP, which may significantly affect mobility, quality of life, and psychological well-being. Although international guidelines, including those of the American College of Obstetricians and Gynecologists (ACOG), recommend physical activity during pregnancy, few interventions specifically target PGP, and the role of pelvic floor function has been largely overlooked.

The pelvic floor contributes to lumbopelvic stability through myofascial connections and motor control. Dysfunction of the pelvic floor muscles is frequently observed in women with PGP, with symptoms such as hypertonicity, poor endurance, and ineffective contractions. Evidence suggests an association between pelvic floor dysfunction and pelvic pain, but no trial to date has combined adapted physical activity with targeted pelvic floor rehabilitation in pregnant women with PGP.

Objectives

The primary objective of this exploratory randomized controlled trial is to evaluate the effect of a combined intervention (adapted physical activity with optional individualized pelvic floor rehabilitation) on pain intensity and functional impact of PGP during pregnancy.

Secondary objectives include:

* To assess the effect of the intervention on pelvic symptoms and pelvic floor functionality.
* To explore the relationship between pelvic floor dysfunction and the course of PGP.
* To evaluate adherence and acceptability of the intervention program.

Study Design

This is a monocentric, randomized, controlled, open-label exploratory trial conducted at Hospital La Tour in Geneva, Switzerland. Forty pregnant women with clinically confirmed PGP will be randomly assigned (1:1) to an intervention group or a control group. Randomization will be stratified by gestational age and baseline pain intensity.

Intervention group: Weekly adapted physical activity sessions in group format (minimum 9 sessions, 60 minutes each), from enrollment until 36-38 weeks of gestation. Sessions alternate between land and pool settings and include lumbopelvic stabilization, core and multifidus strengthening, mobility, and cardiorespiratory training. Women identified with pelvic floor dysfunction at baseline (via the Pelvic Floor Distress Inventory, PFDI-20) will also be offered up to 9 sessions of individualized pelvic floor rehabilitation.

Control group: Standard prenatal follow-up and a flyer with evidence-based recommendations on safe physical activity during pregnancy. No supervised sessions are provided.

Study Population

Eligible participants are pregnant women ≤27 weeks of gestation with clinically confirmed PGP of moderate to severe intensity (VAS ≥3/10). Diagnosis requires typical pain localization and at least 3 positive clinical tests (e.g., P4 test, Patrick FABER, Menell, ASLR). Exclusion criteria include isolated low back pain without pelvic involvement or any medical contraindication to exercise during pregnancy.

Outcomes

1. Primary outcomes:

   * Pain intensity measured by the Visual Analog Scale (VAS, 0-10 cm).
   * Functional impact of PGP measured by the Pelvic Girdle Questionnaire (PGQ, 25 items, score 0-100).
2. Secondary outcomes:

   * Physical activity (Pregnancy Physical Activity Questionnaire, PPAQ).
   * Pelvic symptoms (Pelvic Floor Distress Inventory, PFDI-20).
   * Pelvic floor function (PERFECT scheme by digital palpation).
   * Adherence to intervention (≥75% of sessions attended).
   * Acceptability (post-intervention questionnaire with Likert scales).

Assessments occur at baseline (≤27 weeks), late pregnancy (36-38 weeks), and 3 months postpartum.

Sample Size and Statistical Considerations

Sample size (n=40, 20 per group) was determined based on detecting a clinically meaningful reduction in VAS pain scores, with α=0.05, 95% power, and an expected large effect size (d=0.8). Data will be analyzed on an intention-to-treat basis using descriptive statistics, parametric or non-parametric tests as appropriate, and mixed linear models including relevant covariates (e.g., parity, baseline scores).

Duration and Timeline

The project will last 27 months in total. Enrollment will begin in September 2025 and end in December 2026. The last postpartum follow-up will occur in March 2027, and the study will close in October 2027. Individual participation lasts approximately 6-8 months.

Ethical Considerations

The study is categorized as minimal risk (Category A under Swiss ClinO). All interventions are non-invasive, adapted to pregnancy, and consistent with international standards for prenatal physiotherapy. Approval will be obtained from the Commission Cantonale d'Éthique de la Recherche sur l'être humain (CCER), affiliated with swissethics. Participation is voluntary, and women may withdraw at any time without affecting their standard care. Data will be managed securely in REDCap with strict confidentiality measures.

Significance

This trial will generate new evidence on a comprehensive approach integrating adapted physical activity with pelvic floor rehabilitation for managing pelvic girdle pain in pregnancy. If effective, it could inform physiotherapy practice and contribute to international guidelines, ultimately improving maternal health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥18 years
* Gestational age ≤27 weeks at enrollment
* Clinically confirmed pelvic girdle pain, defined as:
* Pain localized between the posterior iliac crest and the gluteal fold, particularly around the sacroiliac joints and/or pubic symphysis, Pain intensity ≥3/10 on Visual Analog Scale (VAS), At least 3 positive clinical tests among: Posterior Pelvic Pain Provocation (P4) test, Patrick's FABER, Menell's test, Active Straight Leg Raise (ASLR), and palpation of long dorsal sacroiliac ligament or symphysis pubis
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Isolated low back pain without pelvic involvement
* Contraindications to exercise during pregnancy (e.g., severe preeclampsia, placenta previa after 26 weeks, risk of preterm labor, ruptured membranes, significant cardiac or pulmonary disease)
* Neurological, rheumatologic, or orthopedic conditions that may interfere with participation
* Insufficient French language proficiency to understand questionnaires and instructions
* Participation in another interventional study that could affect outcomes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale, VAS) | Baseline (≤27 weeks gestation), 36-38 weeks gestation and 3 months postpartum.
  Pain intensity related to pelvic girdle pain measured on a 10 cm Visual Analog Scale (0 = no pain, 10 = worst imaginable pain).
Functional Impact of Pelvic Girdle Pain (Pelvic Girdle Questionnaire, PGQ) | Baseline, Gestational Weeks 36-38 and 3 months postpartum.
  Functional disability and symptoms assessed with the 25-item Pelvic Girdle Questionnaire (PGQ, score range 0-100; higher scores indicate greater disability).

SECONDARY OUTCOMES:
Physical Activity (Pregnancy Physical Activity Questionnaire, PPAQ) | Baseline, Gestational Weeks 36-38 and 3 months postpartum.
  Self-reported activity levels assessed with the Pregnancy Physical Activity Questionnaire (PPAQ), covering household, occupational, sports/exercise, and transportation domains. Scores reported as MET-hours/week.
Pelvic Symptoms (Pelvic Floor Distress Inventory, PFDI-20) | Baseline, Gestational Weeks 36-38 and 3 months postpartum.
  Pelvic floor symptoms assessed with the 20-item PFDI-20 questionnaire (score range 0-300; higher scores indicate more severe symptoms).
Pelvic Floor Function (PERFECT Scheme) | Baseline and Gestational Weeks 36-38
  Clinical evaluation of pelvic floor muscle function using the PERFECT scheme (Power, Endurance, Repetitions, Fast contractions, Every Contraction Timed), assessed by digital palpation.
Adherence to Intervention | During pregnancy until 36-38 weeks gestation.
  Proportion of participants in the intervention arm who attend ≥75% of scheduled sessions.
Acceptability of Intervention | At 36-38 weeks gestation.
  Participant satisfaction assessed with a post-intervention questionnaire (Likert scale 0-10) regarding the usefulness, feasibility, and comfort of the intervention.

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, no formal plan for IPD sharing has been established. De-identified individual participant data may be made available upon reasonable request to the sponsor (Haute École de Santé Vaud, HESAV) after publication of the main trial results. Any data sharing will require a data sharing agreement and approval by the principal investigator (Professor Jeanne BERTUIT)